CLINICAL TRIAL: NCT01095705
Title: Utility of Hypnosis for Transesophageal Echocardiography
Brief Title: Hypnosis for Transesophageal Echocardiography
Acronym: I-SLEPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P090802; 2009-A01156-51 (Other: IDRCB)
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2010-03

CONDITIONS: Discomfort
Keywords: Hypnosis; Transesophageal Echocardiography; Efficiency of Hypnosis
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional procedure (Active Comparator): Local anaesthesia (Lidocaïne)
  Interventions: Procedure: Conventional procedure
- Conventional procedure + Hypnosis (Experimental): Local anaesthesia (Lidocaïne) and Hypnosis
  Interventions: Procedure: Conventional procedure + Hypnosis

INTERVENTIONS:
Procedure: Conventional procedure — Local anaesthesia (Lidocaïne)
  Arms: Conventional procedure
Procedure: Conventional procedure + Hypnosis — Local anaesthesia (Lidocaïne) + Hypnosis (20 minutes)
  Arms: Conventional procedure + Hypnosis

SUMMARY:
The purpose of this study is to determine the additive value of hypnosis to improve patient comfort during transesophageal echocardiography (TEE).

DETAILED DESCRIPTION:
TEE is a widely used diagnostic test in cardiovascular medicine. However, the test may be a source of discomfort to the patient. Patient intolerance of the echocardiography probe limits the duration of the procedure and therefore its diagnostic success. Current strategies to reduce patient discomfort involve global anesthesia, which carries its own side effects and risks of adverse events. Hypnosis may reduce patient discomfort without impairing alertness. The main goal of this study is to determine the additive value of hypnosis to improve patient comfort during TEE.

ELIGIBILITY:
Inclusion criteria:

* Patient with indication for a Transesophageal Echo (TEE)
* Patient competent to provide written informed consent

Exclusion criteria:

* Patient not subscribed to French Social Security System
* Patient non-French speaking
* Age < 18 years
* Follow-up not possible
* patient declared non competent to give informed consent for the study
* History of severe personality disorder
* Patient with a psychiatric treatment started 30 days before the exam
* Patient pregnant or breast-feeding
* Emergency TEE
* Other indication for general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Level of patient comfort | at Day 0
  Visual Analogic Scale

SECONDARY OUTCOMES:
Rate of procedure failure or non-diagnostic study | at Day 0
Duration of the procedure | at Day 0
Quality of the procedure as assessed by the operator | at Day 0

CONTACTS AND LOCATIONS:
Overall Officials: François TOURNOUX, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital LARIBOISIERE Cardiologie - Laboratoire d'Échocardiographie Doppler, Paris, France